CLINICAL TRIAL: NCT00202852
Title: A Placebo-Controlled, Double-Blinded, Randomized Clinical Trial of Anti-TNF Chimeric Monoclonal Antibody (cA2) in Korean Patients With Active Rheumatoid Arthritis Despite Methotrexate
Brief Title: A Placebo-Controlled, Double-Blinded, Randomized Trial of Remicade in Korean Patients With Rheumatoid Arthritis Despite Methotrexate (Study P04280)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04280
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Other: Placebo; Drug: MTX
- 2 (Experimental)
  Interventions: Biological: Infliximab; Drug: MTX

INTERVENTIONS:
Other: Placebo — Placebo infusions at Weeks 0, 2, and 6 and every 8 weeks through Week 22 + MTX
  Arms: 1
Drug: MTX — Placebo infusions at Weeks 0, 2, and 6 and every 8 weeks through Week 22 + MTX; MTX dose >=12.5 mg/week given orally or parenterally, maximum 20 mg/week
  Arms: 1
Biological: Infliximab — Infliximab 3 mg/kg given as an infusion at Weeks 0, 2, and 6 and every 8 weeks through Week 22 + MTX
  Other Names: Remicade; SCH 215596
  Arms: 2
Drug: MTX — 3 mg/kg infliximab infusions at Weeks 0, 2, and 6 and every 8 weeks through Week 22 + MTX; MTX dose >=12.5 mg/week given orally or parenterally, maximum 20 mg/week
  Arms: 2

SUMMARY:
Prior to the first infusion, patients will be randomized into one of two groups (placebo or infliximab). All patients will continue to receive the same does of methotrexate (MTX) during the study as received prior to the study. The objective of the study is to evaluate the efficacy and safety result of infliximab with Korean patients in reducing clinical signs and symptoms of rheumatoid arthritis (RA) at 30 weeks following the onset of treatment and to review whether the result is comparable to the result of the ATTRACT trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA according to the revised 1987 criteria of the American Rheumatism Association (Arnett et al, 1988). The disease should have been diagnosed at least 6 months prior to screening.
* Active disease at the time of screening and pre-infusion as defined by:

  * >=6 swollen joints
  * >=6 tender joints and 2 of the following:

    * morning stiffness >=45 min
    * ESR >=28 mm/h
    * CRP >=20 mg/L
* Men and women, >=18 to <=75 years of age
* Men and women of childbearing potential must be using adequate birth control measures (abstinence, oral contraceptives, IUD, barrier method with spermicide or, surgical sterilization) and should continue such precautions for 6 months after receiving the last infusion.
* Patients must have been using oral or parenteral MTX for at least 3 months with no break(s) in treatment of more than 2 weeks total during this period. Patients must have been on a stable dose of >=12.5 mg/wk (maximum 20mg/wk) for at least 4 weeks prior to screening.
* Patients must be on a stable dose of folic acid prophylaxis for at least 4 weeks prior to screening.
* Patients using oral corticosteroids, must have been on a stable dose of <=10 mg/day for at least 4 weeks prior to screening. If currently not using corticosteroids the patient must have not received corticosteroids for at least 4 weeks prior to screening.
* If using NSAIDs, patients should have been on a stable dose for at least 4 weeks prior to screening. If currently not using NSAIDs the patient must have been off for at least 4 weeks prior to screening.
* The screening laboratory tests must meet the following criteria:

  * Hemoglobin >=5.3 mmol/L (>=8.5 g/dL), providing a low hemoglobin level is not due to nutritional deficiencies or due to diseases other than chronic RA
  * WBC >=3.5 x 10^9/L
  * Neutrophils >=1.5 x 10^9/L
  * Platelets >=100 x 10^9/L
  * Serum transaminase <=2 times the upper limit of normal
  * Alkaline phosphatase levels <=2 times the upper limit of normal
  * Serum creatinine <=150 µmol/L (<=1.7 mg/dL)
* Patient must be able to adhere to the study visit schedule and other protocol requirements.
* Patient must be capable of giving informed consent and the consent must have been obtained prior to any study procedures including wash-out period.

Exclusion Criteria:

* Pregnant women, nursing mothers or a planned pregnancy within 1.5 years of enrollment.
* Patients who are incapacitated, largely or wholly bedridden or confined to a wheelchair, and who have little or no ability for self-care.
* Patients who have any current systemic inflammatory condition with signs and symptoms that might confound the evaluations of benefit from the Infliximab therapy, eg Lyme disease, or a rheumatic disease other than RA.
* Use of DMARDs other than MTX within 4 weeks prior to screening. (If a patient had prior exposure to leflunomide within the past 6 months, cholestyramine 8 g should be given 3 times daily for 11 days to rapidly lower the plasma level of leflunomide.)
* Use of intra-articular, i.m. or i.v. corticosteroids (including i.m. ACTH) within 4 weeks prior to screening.
* Have been previously treated with infliximab or genetic recombinant therapy with RA (e.g. etanercept, adalimumab).
* Treatment with any other therapeutic agent targeted at reducing TNF (eg, pentoxifylline or thalidomide) within the previous 3 months.
* Treatment with any investigational drug within the previous 3 months.
* Prior use of cyclophosphamide, nitrogen mustard, chlorambucil, or other alkylating agents.
* Have a history of any clinically significant adverse reaction to murine or chimeric proteins, including but not limited to allergic reactions.
* History of infected joint prosthesis within previous 5 years.
* Serious infections, such as hepatitis, pneumonia, pyelonephritis in the previous 3 months.
* Chronic infectious disease such as chronic renal infection, chronic chest infection with bronchiectasis or sinusitis.
* Have active TB. Also excluded are patients who have evidence of latent TB (positive PPD skin test or a history of latent TB) without adequate therapy for TB initiated prior to first infusion of study drug. Also excluded are patients with evidence of an old or latent TB infection without documented adequate therapy, if they will not be treated with antitubercular therapy during the trial. Patients with a current close contact with an individual with active TB will also be excluded. Additionally, patients who have completed treatment for active TB within the previous 2 years are now explicitly excluded from the trial. Patients with a household member who has a history of active pulmonary TB should have had a thorough evaluation for TB prior to study enrollment as recommended by a local infectious disease specialist or published local guidelines of TB control agencies. Also excluded are patients with opportunistic infections, including but not limited to evidence of active cytomegalovirus, active Pneumocystis carinii, aspergillosis, or atypical mycobacterial infection, etc, within the previous 6 months.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic or cerebral disease.
* History of lymphoproliferative disease including lymphoma or signs suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic areas), or splenomegaly.
* Any current known malignancy or history of malignancy within the previous 5 years, except for squamous or basal cell carcinoma of the skin that have been treated with no evidence of recurrence.
* Patients with moderate or severe heart failure (NYHA class III/IV)
* Patients with pre-existing or recent onset of central nervous system demyelinating disorders
* Known recent substance abuse (drug or alcohol).
* Patients in whom multiple venipunctures are not feasible due to poor tolerability or lack of easy access.
* Have a known infection with HIV or known active hepatitis B/C infection (including associated chronic active hepatitis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2005-06-01 (Actual); Primary Completion 2006-03-01 (Actual); Study Completion 2006-03-01 (Actual)

PRIMARY OUTCOMES:
Achievement of a clinical response (according to the ACR criteria) at the 30-week follow-up visit. | 30-week follow-up visit.

SECONDARY OUTCOMES:
Safety evaluations will include measurements of vital signs during and immediately after the infusions of study agents. | During and immediately after the infusions of study agents.
Assessment of adverse events at each of the evaluation visits. | At each evaluation visit.
Routine, laboratory tests (hematology, blood chemistry, and urinalysis) will be performed at Screening, at 2 and 6 weeks, and thereafter every 8 weeks through Week 30 for patients. | At Screening, Week 2, Week 6, and then every 8 weeks thereafter through Week 30.

REFERENCES:
- [Derived] Kim J, Ryu H, Yoo DH, Park SH, Song GG, Park W, Cho CS, Song YW. A clinical trial and extension study of infliximab in Korean patients with active rheumatoid arthritis despite methotrexate treatment. J Korean Med Sci. 2013 Dec;28(12):1716-22. doi: 10.3346/jkms.2013.28.12.1716. Epub 2013 Nov 26. PMID 24339699
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html